CLINICAL TRIAL: NCT04038359
Title: A Phase 2, Randomized, Open-label, 2-Arm Study Comparing 2 Intermittent Dosing Schedules of Duvelisib in Subjects With Indolent Non-Hodgkin Lymphoma (iNHL)
Brief Title: A Phase 2 Study Comparing 2 Intermittent Dosing Schedules of Duvelisib in Participants With Indolent Non-Hodgkin Lymphoma
Acronym: TEMPO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SecuraBio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VS-0145-229; 2019-001381-14 (EudraCT Number)
Record Dates: First submitted 2019-07-10; First posted 2019-07-30 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Indolent Non-Hodgkin Lymphoma
Keywords: PI3K Inhibitor
MeSH Terms: interventions — duvelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Duvelisib, Continuous and Intermittent Dosing (Experimental): Duvelisib 25 milligrams (mg) twice daily (BID) continuously for 10 weeks, followed by 25 mg BID dosed 2 weeks off and 2 weeks on for each subsequent 4-week cycle.
  Interventions: Drug: Duvelisib
- Duvelisib, Intermittent Dosing (Experimental): Duvelisib 25 mg BID dosed 2 weeks on and 2 weeks off.
  Interventions: Drug: Duvelisib

INTERVENTIONS:
Drug: Duvelisib — Phosphoinositide 3-kinase (PI3K) inhibitor
  Other Names: Copiktra; VS-0145; IPI-145

SUMMARY:
This study examined the effects of predefined 2-week duvelisib dose holidays on tumor responses and safety/tolerability.

DETAILED DESCRIPTION:
This was a Phase 2, randomized, open-label, 2-arm study designed to evaluate the efficacy and safety of prescribed drug holidays of duvelisib treatment in participants with relapsed or refractory (R/R) indolent non-Hodgkin lymphoma (iNHL) who have received at least 1 prior systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group performance status ≤ 2
* Histologically confirmed diagnosis of iNHL (subtypes include follicular lymphoma [FL] Grades 1 to 3a), marginal zone lymphoma (splenic, nodal, or extranodal), or small lymphocytic lymphoma
* Must have received 1 prior systemic regimen for iNHL
* Must have documented radiologic evidence of disease progression, at least 1 bi-dimensionally measurable lesion ≥ 1.5 centimeters (which has not been previously irradiated), according to 2007 revised International Working Group criteria, and be a candidate for a subsequent line of therapy.
* Must have adequate organ function defined by the following laboratory parameters:

  * Absolute neutrophil count ≥ 1.0 × 10^9/liter (L)
  * Platelet count ≥ 75 × 10^9/L
  * Hemoglobin ≥ 8 grams/deciliter
  * Estimated creatinine clearance ≥ 60 milliliters/minute, as determined by the Cockcroft-Gault method
  * Total bilirubin ≤ 1.5 × upper limit of normal (ULN) (exception: participants with Gilbert's Syndrome may have a bilirubin > 1.5 × ULN)
  * Aspartate transaminase/serum glutamic-oxaloacetic transaminase and alanine aminotransferase/serum pyruvic transaminase ≤ 3.0 × ULN

Exclusion Criteria:

* Anticancer treatment, major surgery, or use of any investigational drug within 28 days before the start of study intervention; palliative radiation therapy is allowed if > 7 days before planned first dose of study interventions, and any toxicity is Grade ≤ 1
* Clinical or histological evidence of transformation to a more aggressive subtype of lymphoma or grade 3b FL or Richters' transformation or chronic lymphocytic leukemia
* Prior allogeneic hematopoietic stem cell transplant; prior treatment with a PI3K inhibitor
* History of drug-induced colitis or pneumonitis; tuberculosis treatment ≤ 2 years prior to randomization; administration of a live or live attenuated vaccine within 6 weeks of randomization
* Ongoing treatment with chronic immunosuppressants or systemic steroids or treatment for systemic bacterial, fungal, or viral infection
* Active cytomegalovirus or Epstein-Barr virus infection
* Unable to receive prophylactic treatment for pneumocystis, herpes simplex virus, or herpes zoster at screening
* Concurrent administration of medications or foods that are strong inhibitors or inducers of cytochrome P450 3A. No prior use within 2 weeks before the start of study intervention.
* Baseline QT interval corrected with Fridericia's method > 500 milliseconds
* Concurrent active malignancy other than non-melanoma skin cancer or carcinoma in situ of the cervix, bladder cancer, or prostate cancer not requiring treatment. Participants with previous malignancies are eligible if they have been disease-free for 2 years or more.
* Unstable or severe uncontrolled medical condition that would, in the Investigator's judgment, increase the participant's risk to participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-07-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (6):
  - Florida Cancer Specialists - Fort Myers, Fort Myers, Florida
  - Florida Cancer Specialists & Research Institute - Lecanto, Lecanto, Florida
  - Mid-Florida Cancer Centers, Orange City, Florida
  - Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Tennessee Oncology, Nashville, Tennessee
- Czechia (2):
  - FN Hradec Kralove, Hradec Králové
  - Vseobecna fakultni nemocnice v Praze, Prague
- Universitaetsklinikum Bonn AöR, Bonn, Germany
- Italy (5):
  - Oncology Istituto Romagnolo per lo Studio dei Tumori (IRST) Dino Amadori, Meldola, Forli
  - IEO - Istituto Europeo di Oncologia, IRCCS, Milan
  - AUSL di Reggio Emilia IRCCS, Arcispedale Santa Maria Nuova di Reggio Emilia, Reggio Emilia
  - Azienda Ospedaliera Santa Maria di Terni, Terni
  - Ospedale di Circolo, PO Varese, AO Ospedale di Circolo e Fondazione Macchi, Varese
- Poland (3):
  - Wojewodzki Szpital Specjalistyczny im. Janusza Korczaka w Slupsku Sp. z o.o., Słupsk, Pomeranian Voivodeship
  - Pratia Onkologia Katowice, Katowice
  - Centrum Medyczne Pratia Poznan, Skórzewo
- Russia (3):
  - State Budgetary Healthcare Institution of Moscow City Moscow Multidisciplinary Clinical Center "Kommunarka" of the Department of Healthcare of Moscow City, Moscow
  - City Clinical Hospital n.a. Botkin, Moscow
  - First Saint-Petersburg State Medical University n.a. I.P. Pavlov, Saint Petersburg
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center - Oncology, Seoul
  - Samsung Medical Center - Hematology-Oncology, Seoul
- United Kingdom (3):
  - NHS Greater Glasgow & Clyde - CRUK Clinical Trials Unit, Glasgow
  - Royal Liverpool Hospital [Hematology/Transfusion Medicine], Liverpool
  - Christie Hospital NHS Foundation Trust, Manchester

RESULTS

PARTICIPANT FLOW:
Groups:
- Duvelisib, Continuous and Intermittent Dosing: Duvelisib 25 milligrams (mg) twice daily (BID) continuously for 10 weeks, followed by 25 mg BID dosed 2 weeks off and 2 weeks on of each subsequent 4-week cycle.
Period: Overall Study
Arm/Group | Duvelisib, Continuous and Intermittent Dosing | Duvelisib, Intermittent Dosing
Started | 52 | 51
Received At Least 1 Dose of Study Drug (All-treated (AT) Analysis Set/Modified Intent-to-treat (mITT) Analysis Set) | 51 | 51
Completed | 32 | 36
Not Completed | 20 | 15
Not completed — Consent Withdrawn Prior to Receiving Study Drug | 1 | 0
Not completed — Death | 8 | 7
Not completed — Lost to Follow-up | 3 | 0
Not completed — Participant Moved | 1 | 0
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Physician Decision | 3 | 2
Not completed — Adverse Event | 0 | 2
Not completed — Progressive Disease | 0 | 1

BASELINE CHARACTERISTICS:
Population: All-Treated (AT) Analysis Set: All participants who receive at least 1 dose of duvelisib.
Groups:
- Duvelisib, Continuous and Intermittent Dosing: Duvelisib 25 mg BID continuously for 10 weeks, followed by 25 mg BID dosed 2 weeks off and 2 weeks on of each subsequent 4-week cycle.
- Total: Total of all reporting groups
Arm/Group | Duvelisib, Continuous and Intermittent Dosing | Duvelisib, Intermittent Dosing | Total
Number analyzed (Participants) | 51 | 51 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (12.15) | 63.9 (11.40) | 62.2 (11.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 27 | 55
  Male | 23 | 24 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 48 | 50 | 98
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 14 | 9 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 36 | 42 | 78
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) According to the 2007 Revised International Working Group (IWG) Criteria
Description: ORR was defined as the percentage of participants achieving a complete response (CR) or partial response (PR) and assessed using the 2007 revised IWG criteria. The 2007 revised IWG criteria defined CR as the disappearance of all evidence of disease and PR as the regression of measurable disease and no new sites.
Time Frame: Up to 14 months
Population: Modified Intent-to-treat (mITT) analysis set: all participants who receive at least 1 dose of duvelisib. Per-protocol (PP) Analysis Set: all participants in the mITT analysis set who did not violate the protocol in a way that would significantly affect the study outcome. Here, 'Number Analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Duvelisib, Continuous and Intermittent Dosing | Duvelisib, Intermittent Dosing
Number analyzed (Participants) | 49 | 51
percentage of participants
  mITT | 65.3 [50.4 to 78.3] | 52.9 [38.5 to 67.1]
  PP: number analyzed (Participants) | 45 | 46
  PP | 62.2 [46.5 to 76.2] | 54.3 [39.0 to 69.1]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from first dose to first progressive disease (PD) or death (progression date/death date - treatment start date + 1) or, for participants without PD or documented death, as the time from first dose to censoring date (censoring date - treatment start date + 1). The 2007 revised IWG criteria defined PD as any new lesion or increase by ≥50% of previously involved sites from nadir. The 2014 Lugano criteria defined PD as a progressive metabolic response (according to positron emission tomography-computed tomography [PET-CT]) and progressive disease (according to computed tomography [CT]). Results reported as months.
Time Frame: Up to 2 years
Population: Modified Intent-to-treat (mITT) analysis set: all participants who receive at least 1 dose of duvelisib. Here, 'Overall Number of Participants Analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Duvelisib, Continuous and Intermittent Dosing | Duvelisib, Intermittent Dosing
Number analyzed (Participants) | 49 | 51
months
  2007 Revised IWG Criteria | 16.0 [8.5 to 27.2] | 23.0 [12.5 to 34.3]
  2014 Lugano Criteria | 16.0 [8.5 to 27.2] | 23.0 [12.5 to 34.3]

3. Secondary Outcome: ORR At Specific Timepoints
Description: ORR at 6, 12, 18, and 24 months after first dose of study intervention was defined as the percentage of participants achieving CR or PR at each timepoint and was assessed using both the 2007 revised IWG criteria and the 2014 Lugano criteria. The 2007 revised IWG criteria defined CR as the disappearance of all evidence of disease and PR as the regression of measurable disease and no new sites. The 2014 Lugano criteria defined CR as a complete metabolic response (according to PET-CT) and a complete radiologic response (according to CT) and PR as partial metabolic response (according to PET-CT) and partial remission (according to CT). The response was cumulative for each timepoint; a participant was considered a responder if their first response occurred up to the end of that timepoint.
Time Frame: 6, 12, 18, and 24 months after first dose of study intervention
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Duvelisib, Continuous and Intermittent Dosing | Duvelisib, Intermittent Dosing
Number analyzed (Participants) | 49 | 51
percentage of participants
  6 months: 2007 Revised IWG Criteria | 63.3 [48.3 to 76.6] | 49.0 [34.8 to 63.4]
  12 months: 2007 Revised IWG Criteria | 65.3 [50.4 to 78.3] | 52.9 [38.5 to 67.1]
  18 months: 2007 Revised IWG Criteria | 65.3 [50.4 to 78.3] | 52.9 [38.5 to 67.1]
  24 months: 2007 Revised IWG Criteria | 65.3 [50.4 to 78.3] | 52.9 [38.5 to 67.1]
  6 months: 2014 Lugano Criteria | 63.3 [48.3 to 76.6] | 47.1 [32.9 to 61.5]
  12 months: 2014 Lugano Criteria | 65.3 [50.4 to 78.3] | 51.0 [36.6 to 65.2]
  18 months: 2014 Lugano Criteria | 65.3 [50.4 to 78.3] | 51.0 [36.6 to 65.2]
  24 months: 2014 Lugano Criteria | 65.3 [50.4 to 78.3] | 51.0 [36.6 to 65.2]

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined for participants with CR or PR as the time from the date of first documentation of response (CR or PR) to date of the first documentation of PD or death. The 2007 revised IWG criteria defined CR as the disappearance of all evidence of disease, PR as the regression of measurable disease and no new sites, and PD as any new lesion or increase by ≥50% of previously involved sites from nadir. The 2014 Lugano criteria defined CR as a complete metabolic response (according to PET-CT) and a complete radiologic response (according to CT), PR as partial metabolic response (according to PET-CT) and partial remission (according to CT), and PD as a progressive metabolic response (according to PET-CT) and progressive disease (according to CT). Results are reported as months.
Time Frame: Up to 2 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Duvelisib, Continuous and Intermittent Dosing | Duvelisib, Intermittent Dosing
Number analyzed (Participants) | 49 | 51
months
  2007 Revised IWG Criteria | 21.4 [13.7 to NA] — Insufficient number of participants with events. | 32.2 [17.5 to NA] — Insufficient number of participants with events.
  2014 Lugano Criteria | 21.4 [13.7 to NA] — Insufficient number of participants with events. | 32.2 [13.8 to NA] — Insufficient number of participants with events.

5. Secondary Outcome: Overall Survival (OS)
Description: OS was the time from first dose to death (death date - treatment start date + 1). Participants without documented death were censored at their last known alive date (last known alive date - treatment start date + 1). Results reported as months.
Time Frame: Up to 2 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Duvelisib, Continuous and Intermittent Dosing | Duvelisib, Intermittent Dosing
Number analyzed (Participants) | 49 | 51
months | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events.

6. Secondary Outcome: Lymph Node Response Rate (LNRR)
Description: LNRR was calculated as the percentage of participants achieving ≥50% decrease in the sum of the product of the diameters of target lymph nodes. The confidence interval for LNRR was calculated only for participants who had at least 1 nodal target lesion, using the Clopper-Pearson exact method for binomial proportions. Participants whose target lesions were all extranodal were excluded from this analysis.
Time Frame: 14 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Duvelisib, Continuous and Intermittent Dosing | Duvelisib, Intermittent Dosing
Number analyzed (Participants) | 49 | 51
percentage of participants | 64.3 [48.0 to 78.4] | 60.9 [45.4 to 74.9]

7. Secondary Outcome: Time To First Response (TTFR)
Description: For participants with CR or PR, TTFR was defined as the time from first dose of study intervention to time of first CR or PR and was calculated as: the date of first CR or PR - randomization date + 1. The 2007 revised IWG criteria defined CR as the disappearance of all evidence of disease and PR as the regression of measurable disease and no new sites. The 2014 Lugano criteria defined CR as a complete metabolic response (according to PET-CT) and a complete radiologic response (according to CT) and PR as partial metabolic response (according to PET-CT) and partial remission (according to CT). Results are reported as months.
Time Frame: Up to 14 months
Population: Modified Intent-to-treat (mITT) analysis set: all participants who receive at least 1 dose of duvelisib. Here, 'Number Analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: months
Arm/Group | Duvelisib, Continuous and Intermittent Dosing | Duvelisib, Intermittent Dosing
Number analyzed (Participants) | 49 | 51
months
  2007 Revised IWG Criteria: number analyzed (Participants) | 32 | 27
  2007 Revised IWG Criteria | 2.30 [2.1 to 12.9] | 2.30 [2.1 to 12.5]
  2014 Lugano Criteria: number analyzed (Participants) | 32 | 26
  2014 Lugano Criteria | 2.30 [2.1 to 12.9] | 2.30 [2.1 to 12.5]

8. Secondary Outcome: Time To Treatment Failure (TTF)
Description: TTF was calculated as the time from first dose of study treatment to discontinuation for any reason (discontinuation date - treatment start date + 1). Participants who were still ongoing treatment at time of data cut were censored (last dose date - treatment start date + 1). Results reported as months.
Time Frame: Up to 2 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Duvelisib, Continuous and Intermittent Dosing | Duvelisib, Intermittent Dosing
Number analyzed (Participants) | 49 | 51
months | 12.6 [6.2 to 17.1] | 14.3 [8.0 to 23.0]

9. Secondary Outcome: ORR According to 2014 Lugano Criteria
Description: ORR was defined as the percentage of participants achieving a CR or PR and was assessed using the 2014 Lugano criteria. The 2014 Lugano criteria defined CR as a complete metabolic response (according to PET-CT) and a complete radiologic response (according to CT) and PR as partial metabolic response (according to PET-CT) and partial remission (according to CT).
Time Frame: Up to 14 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Duvelisib, Continuous and Intermittent Dosing | Duvelisib, Intermittent Dosing
Number analyzed (Participants) | 49 | 51
percentage of participants
  mITT | 65.3 [50.4 to 78.3] | 51.0 [36.6 to 65.2]
  PP: number analyzed (Participants) | 45 | 46
  PP | 62.2 [46.5 to 76.2] | 52.2 [36.9 to 67.1]

ADVERSE EVENTS:
Time Frame: Up to 37 months
Description: All reported safety data based upon All-treated Analysis Set: all participants who receive at least 1 dose of duvelisib.
Arm/Group | Duvelisib, Continuous and Intermittent Dosing | Duvelisib, Intermittent Dosing
All-Cause Mortality (participants affected / at risk) | 8/51 | 7/51
Serious Adverse Events (participants affected / at risk) | 13/51 | 16/51
Other Adverse Events (participants affected / at risk) | 49/51 | 50/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duvelisib, Continuous and Intermittent Dosing (N=51) | Duvelisib, Intermittent Dosing (N=51)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Pylorospasm (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Disease progression (General disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 3 | 3
COVID-19 (Infections and infestations) | 2 | 1
Cellulitis (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Major depression (Psychiatric disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 0
Pelvic venous thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Duvelisib, Continuous and Intermittent Dosing (N=51) | Duvelisib, Intermittent Dosing (N=51)
Anaemia (Blood and lymphatic system disorders) | 4 | 5
Neutropenia (Blood and lymphatic system disorders) | 10 | 17
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 4 | 2
Constipation (Gastrointestinal disorders) | 6 | 3
Diarrhoea (Gastrointestinal disorders) | 17 | 10
Dyspepsia (Gastrointestinal disorders) | 5 | 3
Nausea (Gastrointestinal disorders) | 7 | 8
Stomatitis (Gastrointestinal disorders) | 3 | 4
Vomiting (Gastrointestinal disorders) | 5 | 1
Asthenia (General disorders) | 6 | 1
Fatigue (General disorders) | 7 | 5
Pyrexia (General disorders) | 9 | 9
COVID-19 (Infections and infestations) | 8 | 10
Pneumonia (Infections and infestations) | 2 | 5
Upper respiratory tract infection (Infections and infestations) | 4 | 3
Urinary tract infection (Infections and infestations) | 5 | 2
Alanine aminotransferase increased (Investigations) | 15 | 8
Aspartate aminotransferase increased (Investigations) | 15 | 6
Neutrophil count decreased (Investigations) | 3 | 2
Platelet count decreased (Investigations) | 3 | 2
Weight decreased (Investigations) | 3 | 4
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 4
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Dizziness (Nervous system disorders) | 2 | 3
Headache (Nervous system disorders) | 8 | 1
Insomnia (Psychiatric disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 4
Rash (Skin and subcutaneous tissue disorders) | 4 | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 2
Hypertension (Vascular disorders) | 0 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/59/NCT04038359/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-31): https://cdn.clinicaltrials.gov/large-docs/59/NCT04038359/SAP_001.pdf